CLINICAL TRIAL: NCT06828328
Title: A Phase I Study of Engineered Tumor Infiltrating Lymphocytes Injection (GC203 TIL) in Patients With Pancreatic Ductal Adenocarcinoma
Brief Title: A Study of GC203 TIL in PDCA (RJ)
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Juncell Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC203-2024-RJ-PDCA
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-02

CONDITIONS: Pancreatic Cancer; Pancratic Ductal Adenocarcinoma; Treatment Side Effects; Tumor Infiltrating Lymphocytes
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GC203 TIL (Experimental): 5x10^8-1.5x10^10 ±20% in vitro expanded GC203 TILs will be infused i.v. to patients with pancreatic ductal adenocarcinoma after NMA lymphodepletion treatment with hydroxychloroquine(600mg,single-dose) and cyclophosphamide.
  Interventions: Biological: GC203 TIL

INTERVENTIONS:
Biological: GC203 TIL — the candidates will be assigned to GC203 TIL(gene-edited TIL) group

SUMMARY:
This study is to investigate the safety and efficacy of gene-edited tumor infiltrating lymphocyte (GC203 TIL) therapy in patients with pancreatic ductal adenocarcinoma. Gene-edited TILs are expanded from tumor resections or biopsies and infused i.v. into the patient after NMA lymphodepletion treatment with hydroxychloroquine(600mg,single-dose) and cyclophosphamide.

ELIGIBILITY:
Inclusion Criteria:

1. have done the tumor resection for gene-edited GC203 TIL production and successfully produced；
2. Age: 18 years to 70 years;
3. Histologically diagnosed as pancreatic ductal adenocarcinoma;
4. Expected life-span more than 3 months;
5. ECOG score 0-1;
6. Test subjects have failed standard treatment regimens, and be willing to recieve gene-edited GC203 TIL therapy;
7. At least 1 evaluable tumor lesion;
8. Hematology and Chemistry（within 7 days prior to enrollment）:

Absolute count of white blood cells≥2.5×10^9/L; Absolute count of neutropils≥1.5×10^9/L; Absolute count of lymphocytes ≥0.7×109/L； Platelet count≥90×10^9； hemoglobin≥90 g/L; Activated partial thromboplastin time (APTT) ≤1.5xULN (Unless received anticoagulant therapy within the previous 3 days); International normalized ratio (INR) ≤1.5xULN (Unless received anticoagulant therapy within the previous 3 days); Serum creatinine ≤1.5mg/dL(or ≤132.6μmol/L), or clearance rate≥50mL/min; Serum ALT/AST ≤3×ULN(subjects with liver metastasis ≤3×ULN); Totol bilirubin≤1.5×ULN; 9.Test subjects with child-bearing potential must be willing to practice approved highly effective methods of contraception at the time of informed consent, and continue within 1 year after the completion of lymphodepletion； 10.Any malignant tumor-targeting therapies, including radiotherapy, chemotherapy and biologics must cease 28 days before obtaining TILs; 12.Be able to understand and sign the informed consent document; 13.Be able to stick to follow-up visit plan and other requirements in the agreement.

Exclusion Criteria:

1. with other malignant tumors,except for the malignancies that have been cured, have been inactive for ≥5 years prior to study inclusion and have a very low risk of recurrence; Non-melanoma skin cancer or malignant lentigo with adequate treatment and no evidence of disease recurrence; Carcinoma in situ with adequate treatment and no evidence of disease recurrence;
2. Need glucocorticoid treatment, and daily dose of Prednisone greater than 10mg(or equivalent doses of hormones) or outoimmune diseases requiring immunomodulatory treatment;
3. Breathe indoor air in a quiet state, and the oxygen saturation of finger pulse is < 95%;
4. Human immunodeficiency virus (HIV) infection or anti-HIV antibody positive, active HBV or HCV infection (HBsAg positive and/or anti-HCV positive), syphilis infection or Treponema pallidum antibody positive;
5. Significant cardiovascular anomalies according to any of the following definition:

   New York Heart Association (NYHA) Grade III or IV congestive heart failure, clinically significant low blood pressure, uncontrollable symptomatic coronary artery diseases, or ejection fraction less than 35%; Severe cardiac rhythm and conduction anomaly, such as ventricular arrhythmia requiring clinical intervention, second-third degree atrio-ventricular conductive block, etc.
6. Uncontrolled metabolic disorders, such as diabetes, which is known to be uncontrolled, or other non-malignant organ or systemic disease or cancer secondary reactions, can lead to higher medical risk and/or uncertainty in the evaluation of survival;
7. Patients with esophageal or gastric varices requiring immediate intervention (e.g., ligation or sclerotherapy) or who, in the opinion of the investigator or in consultation with a gastroenterologist or hepatologist, have evidence of portal hypertension (including splenomegalgia on imaging) or a history of varicose bleeding must undergo endoscopic evaluation within the first 3 months of enrollment;
8. Hepatic encephalopathy, hepatorenal syndrome or Child-Pugh grade B or more severe cirrhosis, liver failure;
9. Pulmonary fibrosis, interstitial lung disease (both past and present), acute lung disease;
10. Clinically uncontrollable third space effusion, such as pleural fluid and ascites that could not be controlled by drainage or other means prior to enrollment;
11. Patients with known pnelmeningeal metastases; Other patients known to have uncontrolled or untreated central nervous system metastases that are not effectively controlled by treatment, except those who have been treated and whose symptoms are stable, and who discontinue glucocorticoid and anticonvulsant therapy ≥4 weeks prior to cell retransfusion;
12. Severe physical or mental diseases;
13. Have a systemic active infection requiring treatment, or have positive blood cultures(or imaging evidence of infection);
14. Having been treated within a month or being treated now with other medicines, or other biologic therapy, chemo-or radiotherapy;
15. History of allogeneic T cell therapy;
16. Having received immunotherapy and developed irAE level greater than Level 3;
17. Previous anti-tumor treatment AE did not return to CTCAE5.0 version grade 1 or below (toxicity considered by the investigator as non-safety concerns like alopecia excluded);
18. Females in pregnancy or lactation;
19. History of organ transplantation, allogeneic stem cell transplantation, and renal replacement therapy;
20. Researchers considering the test subject as having a history of other severe systemic diseases, or other reasons inappropriate for the clinical study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 6 months
  To characterize the safety profile of GC203 TIL in patients with pancreatic ductal adenocarcinoma who were failed to standard treatment as assessed by incidence of adverse events.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 36 months
  Proportion of patients with response per Response Evaluation Criteria in Solid Tumors (RECIST v1.1)
Disease Control Rate (DCR） | Up to 36 months
  Percentage of patients that meet CR, PR and SD criteria set in this study according to RECIST 1.1
Duration of Response (DOR) | Up to 36 months
  The time length between the first confirmed objective response per RECIST 1.1 to the treatment and the subsequent disease progression per RECIST 1.1
Progression-Free Survival (PFS) | Up to 36 months
  The time length between TIL infusion and confirmed subsequent disease progression according to RECIST 1.1
Overall Survival(OS) | Up to 36 months
  The time length between TIL infusion and death

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes